CLINICAL TRIAL: NCT03406494
Title: Southern Medical University Clinical Research Project Initiative：Efficacy and Safety of a Multicomponent Physical Therapy Program in Mechanically Ventilated Patient With Sepsis
Brief Title: Efficacy and Safety of a Multicomponent Physical Therapy Program in Mechanically Ventilated Patient With Sepsis
Acronym: PTMVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Wang Hua, Vice Director of Critical Care Department, Zhujiang Hospital, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LC2016PY036
Record Dates: First submitted 2017-12-25; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Sepsis
Keywords: sepsis; critical illness; intensive care unit; mechanical ventilation; rehabilitation; mortality; physical function; health-related quality of life
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, assessor-blinded, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be independent from the study and blinded from patient allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Early multicomponent physical therapy program plus sepsis standard therapy
  Interventions: Other: Early multicomponent physical therapy program
- control group (No Intervention): Sepsis standard therapy, including early initiation of intravenous antibiotics, infection source debriding, appropriate fluid therapy, minimum sedation, protocolized weaning procedure, blood glucose control and early enteral feeding, etc.

INTERVENTIONS:
Other: Early multicomponent physical therapy program — 1. Positioning (upright bed standing; turning, moving on bed).
  2. Peripheral muscle strength training (active or passive full range of motion, lower extremities ergometer cycling).
  3. Respiratory muscle training (supine abdominal breathing training).
  4. Neuromuscular electrical stimulation (NMES) on target muscles (bilateral bicipital muscles, quadriceps femoris muscles and rectus femoris).
  5. Gut rehabilitation (midfrequency NMES; abdominal manual or vibration massage).
  Arms: intervention group

SUMMARY:
Despite of a remarkable decrease in overall mortality has been achieved following the International Guidelines for Management of Sepsis and Septic Shock since 2004,the short-and long-term outcomes remain poor in critically ill sepsis patients who had experienced prolonged ventilation in the Intensive Care Unit (ICU). The reason could be due to some subsequent complications developed in the ICU rather than original disease, e.g., ICU-acquired weakness (ICUAW), delirium, diaphragmatic dysfunction (DD) and acute gastrointestinal (GI) injury, which are still not fully recognized or dealt with in a majority of ICU settings across China. This study is aimed to examine whether a multi-component physical therapy (PT) program against these lethal ICU-related complications could reduce ICU 28-day mortality, improve independent functional status and 1-year survival in this subset of patients.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, assessor-blinded, randomized controlled trial and will be conducted in 9 medical ICUs at 7 tertiary hospitals in Southern China. Mechanically ventilated septic patient admitted into ICU will be screened for eligibility into the study. When medically stable, patients randomize into the intervention group will receive a multi-component PT. The PT program is designed to counteract ICUAW, delirium, DD and acute GI injury, and consists of 5 consecutive sessions including positioning, extremities muscle strength training, respiratory muscle strength training, neuromuscular electrical stimulation (NMES) and gut rehabilitation. Each PT session will last for 30 minutes and be provided once daily, 5 days per week, and tailored for each individual subject. PT intervention will continue throughout patient's ICU stay or the primary endpoint is reached. The primary outcome will be the ICU 28-day all-cause mortality, and the secondary outcome measures, e.g., incidences or duration of ICUAW, delirium, DD and acute GI injury, mechanical ventilation outcomes (ventilator dependence, ventilator-free days), adverse events, restoration to independent functional status and long-term survival, will be assessed at preset time points of interviews during periods of treatment and 1-year follow-up after discharge from hospital. The total in-hospital and re-hospitalization costs in the intervention group will be also analyzed and compared to control group to assess the cost-effectiveness of the rehabilitation program.To our knowledge, this study is the first randomized controlled trial examining the efficacy and safety of a multi-component PT program in critically ill sepsis patients on ventilator. Given that rehabilitation is not a routine therapy across most ICUs in China, If this PT program is found to be of mortality benefit, it will provide an alternative non-pharmaceutical approach to deal with these lethal ICU-related complications and reduce the subsequent death. It will also provide useful information for clinical decision and local medical policies making, as well as identifying sepsis patient population who might best benefit from early rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with sepsis in accordance with the Sepsis-3 Criteria.
2. 16 ≤ age ≤ 75 years.
3. Mechanically ventilated for less than 72 hours at recruitment and expected to continue for at least 3 days.
4. Ability to obtain informed consent from patient or proxy.

Exclusion Criteria:

1. acute central nervous system disease (e.g. severe cerebral injury, acute cerebral hemorrhage, brain infarction).
2. active neuromuscular diseases that limiting patient to physical training (e.g. amyotrophic lateral sclerosis, multiple sclerosis, myasthenia gravis, polymyositis, muscular dystrophy).
3. severe thoracic or abdominal trauma.
4. acute myocardial infarction, severe arrhythmia, acute heart failure, hemo-dynamic instability or shock.
5. drug abuse, alcohol addiction, opiates or other drug dependence and psychiatric disorder history.
6. known pregnancy.
7. malignant tumor, cachexia, end stage of chronic illness.
8. contraindications to rehabilitation therapy.
9. inability to obtain an informed consent from patient or a proxy.
10. any other factors such as fractures or limb malformation, that would prevent response to physical exercise or cause injury to the patient.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
ICU 28-day mortality | Through 28-day study period in the ICU.
  Sepsis or non-sepsis related death, undetermined cause of death.

SECONDARY OUTCOMES:
Incidence of ICU-required weakness | Assessed on the day of recruitment, repeated on the days of first try to wean from ventilator, ICU discharge and hospital discharge, with an average of 1 month.
  Using the Medical Research Council (MRC) Score for Muscle Strength to test 12 muscle groups in upper extremities (wrist flexion, elbow flexion, shoulder abduction) and lower extremities (dorsiflexion, knee extension, hip flexion). The MRC sum score ranges from 0 (complete paralysis) to 60 (full strength) as determined by manual muscle testing (MMT), which grades muscle strength from 0 (paralysis) to 5 (normal muscle strength) in each muscle group tested. Patient with a MRC sum score of < 48 or a mean MRC score of < 4 per muscle group will be considered to have ICUAW. If measurement is impossible at recruitment, patient will be deemed as without ICUAW by a Barthel Index score > 60, which ranges from 0 (complete dependence) to 100 (complete independence), collected from a proxy reflecting baseline independent functional status 2 weeks prior to critical illness.
Incidence of delirium | Assessed on the day of recruitment, repeated on the days of first try to wean from ventilator, ICU discharge and hospital discharge, with an average of 1 month.
  Acute cerebral dysfunction with altered mental status, inattention, and either disordered thinking or an altered level of consciousness as determined by the Confusion Assessment Method for the ICU (CAM-ICU). If assessment is impossible at recruitment, patient will be considered without delirium by absence of a history of insanity collected from a proxy reflecting baseline mental status 2 weeks prior to critical illness.
Incidence of diaphragmatic dysfunction | Assessed on the day of first try to wean from ventilator, repeated on the days of ICU discharge and hospital discharge, with an average of 1 month.
  Maximum negative inspiratory pressure (PImax) less than - 80 cm H2O is usually considered to have clinically important inspiratory muscle weakness. Measurements will be performed by using inspiratory hold key on ventilator (intubated patient) or a one-way exhalation valve placed on the opening of mouth (extubated patient). Patient will be instructed to perform maximal inspiratory efforts for 20 seconds against occluded airway at functional residual lung volume (FRC), and change in pressure be recorded by an external data acquisition system (Powerlab/16sp ML795, Australia ADInstruments) through a physiological pressure sensor (MLT 844, Australia ADInstruments) connected to the opening of endotracheal tube or the valve. The signal sampling frequency will be set at 100 Hz and low-pass filtering frequency at 20 Hz. The signal collected will be digitalized and analyzed in a manner of time-domain, and the PImax be recorded after 3 repetitions.
Incidence of acute gastrointestinal injury | Assessed on the day of recruitment, repeated on the days of first try to wean from ventilator, ICU discharge and hospital discharge, with an average of 1 month.
  Malfunctioning of the GI tract in critically ill patients due to their acute illness, distinguished and graded by severity of GI symptoms (e.g., feeding intolerance, vomiting, diarrhoea, paralysis, high gastric residual volumes (HGRVs). Acute gastrointestinal injury (AGI) grade I: increased risk to develop GI dysfunction or failure; AGI grade II: GI dysfunction (interventions required); AGI grade III: GI failure (GI function cannot be restored with interventions); AGI grade IV: dramatically manifesting GI failure.
Ventilator dependence | Number of days required to weaning after the first try, number of days on ventilator, assessed within an average of 3 weeks.
  Referred to one of the following categories: difficult weaning: fail initial weaning and require up to 3 spontaneous breath test (SBT) or ≤7 days to achieve success; delayed weaning: fail at least 3 weaning attempts or require > 7 days to weaning after the first SBT; prolonged mechanical ventilation (PMV): requiring ventilator support for more than 21 days.
Adverse events | Through physical therapy periods, an average of 1 month.
  Unexpected physiologic response or patient complaints to physical exercise, e.g., more than 20% variability in rest heart rate; 110 mmHg < mean arterial pressure < 60 mmHg; decremental pulse oximetry < 90%; severe dyspnea as determined by the Modified Borg Dyspnea Scale > 4 (ranged from 0-10, indicative of dyspnea degree from just noticeable to maximum); patient-ventilator asynchrony; altered mentation; catheters or tubes displacement; documented organ damage; accidental death.
Length of stay | From admission to ICU discharge and hospital discharge, estimated between 4 to 6 weeks.
  Number of days spent in the ICU or hospital.
Independent functional status | The 3rd, 6th and 12th months of 1-year follow up after hospital discharge.
  Referred to ability to perform 10 activities of daily living (ADL's), including eating, transfer from bed to chair, dressing, toileting, bathing, grooming, walking, stair climbing, maintaining continence. Independent functional status is determined by a Barthel Index Score > 60, which ranged from 0 (complete dependence) to 100 (complete independence).
Health-related quality of life (HRQOL) | The 3rd, 6th and 12th months of 1-year follow up after hospital discharge.
  Evaluated by using the mandarin version Short-Form-36 Questionnaire translated by the Zhejiang University, China., consisting of eight domains (e.g., physical function (PF), role limitations due to physical problems (RP), body pain (BP), general health (GH), vitality (VT), social function (SF), role limitations due to emotional problems (RE), mental health (MH). The combined score for each domain is obtained by summing score of each item contained in the domain and directly converted into a 0-100 score scale using the Likert method of summated ratings. A score scale of zero is equivalent to maximum disability and 100 equals to the best possible health state.
One-year mortality | One year.
  All-cause death during 1-year follow-up after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, Study Director — Zhujiang Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Zhang SW, Wang H, Su Q, Wang BE, Wang C, Yin CH; MODS Research Group. [Clinical epidemiology of 1,087 patients with multiple organ dysfunction syndrome]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2007 Jan;19(1):2-6. Chinese. PMID 17207352
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM; Surviving Sepsis Campaign Management Guidelines Committee. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Crit Care Med. 2004 Mar;32(3):858-73. doi: 10.1097/01.ccm.0000117317.18092.e4. PMID 15090974
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Murphy CV, Schramm GE, Doherty JA, Reichley RM, Gajic O, Afessa B, Micek ST, Kollef MH. The importance of fluid management in acute lung injury secondary to septic shock. Chest. 2009 Jul;136(1):102-109. doi: 10.1378/chest.08-2706. Epub 2009 Mar 24. PMID 19318675
- [Background] Zhou J, Tian H, Du X, Xi X, An Y, Duan M, Weng L, Du B; for China Critical Care Clinical Trials Group (CCCCTG). Population-Based Epidemiology of Sepsis in a Subdistrict of Beijing. Crit Care Med. 2017 Jul;45(7):1168-1176. doi: 10.1097/CCM.0000000000002414. PMID 28422777
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] MacIntyre NR. The ventilator discontinuation process: an expanding evidence base. Respir Care. 2013 Jun;58(6):1074-86. doi: 10.4187/respcare.02284. PMID 23709201
- [Background] Thille AW, Cortes-Puch I, Esteban A. Weaning from the ventilator and extubation in ICU. Curr Opin Crit Care. 2013 Feb;19(1):57-64. doi: 10.1097/MCC.0b013e32835c5095. PMID 23235542
- [Background] Chang AT, Boots RJ, Brown MG, Paratz J, Hodges PW. Reduced inspiratory muscle endurance following successful weaning from prolonged mechanical ventilation. Chest. 2005 Aug;128(2):553-9. doi: 10.1378/chest.128.2.553. PMID 16100137
- [Background] Vincent JL, Shehabi Y, Walsh TS, Pandharipande PP, Ball JA, Spronk P, Longrois D, Strom T, Conti G, Funk GC, Badenes R, Mantz J, Spies C, Takala J. Comfort and patient-centred care without excessive sedation: the eCASH concept. Intensive Care Med. 2016 Jun;42(6):962-71. doi: 10.1007/s00134-016-4297-4. Epub 2016 Apr 13. PMID 27075762
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Schweickert WD, Hall J. ICU-acquired weakness. Chest. 2007 May;131(5):1541-9. doi: 10.1378/chest.06-2065. PMID 17494803
- [Background] Trogrlic Z, van der Jagt M, Bakker J, Balas MC, Ely EW, van der Voort PH, Ista E. A systematic review of implementation strategies for assessment, prevention, and management of ICU delirium and their effect on clinical outcomes. Crit Care. 2015 Apr 9;19(1):157. doi: 10.1186/s13054-015-0886-9. PMID 25888230
- [Background] Leslie DL, Inouye SK. The importance of delirium: economic and societal costs. J Am Geriatr Soc. 2011 Nov;59 Suppl 2(Suppl 2):S241-3. doi: 10.1111/j.1532-5415.2011.03671.x. PMID 22091567
- [Background] Skrobik Y. Delirium prevention and treatment. Crit Care Clin. 2009 Jul;25(3):585-91, x. doi: 10.1016/j.ccc.2009.05.003. PMID 19576532
- [Background] Wang JY, Wu H, Tong ZD, Yan JB, Li KF, Tang A. [A review on the epidemiologic features of severe fever with thrombocytopenia syndrome]. Zhonghua Liu Xing Bing Xue Za Zhi. 2016 Feb;37(2):294-8. doi: 10.3760/cma.j.issn.0254-6450.2016.02.029. Chinese. PMID 26917534
- [Background] Reintam Blaser A, Malbrain ML, Starkopf J, Fruhwald S, Jakob SM, De Waele J, Braun JP, Poeze M, Spies C. Gastrointestinal function in intensive care patients: terminology, definitions and management. Recommendations of the ESICM Working Group on Abdominal Problems. Intensive Care Med. 2012 Mar;38(3):384-94. doi: 10.1007/s00134-011-2459-y. Epub 2012 Feb 7. PMID 22310869
- [Background] Laghi F, Cattapan SE, Jubran A, Parthasarathy S, Warshawsky P, Choi YS, Tobin MJ. Is weaning failure caused by low-frequency fatigue of the diaphragm? Am J Respir Crit Care Med. 2003 Jan 15;167(2):120-7. doi: 10.1164/rccm.200210-1246OC. Epub 2002 Oct 31. PMID 12411288
- [Background] Hermans G, Agten A, Testelmans D, Decramer M, Gayan-Ramirez G. Increased duration of mechanical ventilation is associated with decreased diaphragmatic force: a prospective observational study. Crit Care. 2010;14(4):R127. doi: 10.1186/cc9094. Epub 2010 Jul 1. PMID 20594319
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Garnacho-Montero J, Madrazo-Osuna J, Garcia-Garmendia JL, Ortiz-Leyba C, Jimenez-Jimenez FJ, Barrero-Almodovar A, Garnacho-Montero MC, Moyano-Del-Estad MR. Critical illness polyneuropathy: risk factors and clinical consequences. A cohort study in septic patients. Intensive Care Med. 2001 Aug;27(8):1288-96. doi: 10.1007/s001340101009. PMID 11511941
- [Background] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Background] Supinski GS, Callahan LA. Diaphragm weakness in mechanically ventilated critically ill patients. Crit Care. 2013 Jun 20;17(3):R120. doi: 10.1186/cc12792. PMID 23786764
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Jul 17;371(3):287-8. doi: 10.1056/NEJMc1406274. No abstract available. PMID 25014703
- [Background] Hermans G, De Jonghe B, Bruyninckx F, Van den Berghe G. Interventions for preventing critical illness polyneuropathy and critical illness myopathy. Cochrane Database Syst Rev. 2014 Jan 30;2014(1):CD006832. doi: 10.1002/14651858.CD006832.pub3. PMID 24477672
- [Background] Petrof BJ, Jaber S, Matecki S. Ventilator-induced diaphragmatic dysfunction. Curr Opin Crit Care. 2010 Feb;16(1):19-25. doi: 10.1097/MCC.0b013e328334b166. PMID 19935062
- [Background] Ayas NT, McCool FD, Gore R, Lieberman SL, Brown R. Prevention of human diaphragm atrophy with short periods of electrical stimulation. Am J Respir Crit Care Med. 1999 Jun;159(6):2018-20. doi: 10.1164/ajrccm.159.6.9806147. PMID 10351955
- [Background] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346
- [Background] Smith BK, Gabrielli A, Davenport PW, Martin AD. Effect of training on inspiratory load compensation in weaned and unweaned mechanically ventilated ICU patients. Respir Care. 2014 Jan;59(1):22-31. doi: 10.4187/respcare.02053. Epub 2013 Jun 13. PMID 23764858
- [Background] Doig GS, Heighes PT, Simpson F, Sweetman EA. Early enteral nutrition reduces mortality in trauma patients requiring intensive care: a meta-analysis of randomised controlled trials. Injury. 2011 Jan;42(1):50-6. doi: 10.1016/j.injury.2010.06.008. PMID 20619408
- [Background] Balas MC, Burke WJ, Gannon D, Cohen MZ, Colburn L, Bevil C, Franz D, Olsen KM, Ely EW, Vasilevskis EE. Implementing the awakening and breathing coordination, delirium monitoring/management, and early exercise/mobility bundle into everyday care: opportunities, challenges, and lessons learned for implementing the ICU Pain, Agitation, and Delirium Guidelines. Crit Care Med. 2013 Sep;41(9 Suppl 1):S116-27. doi: 10.1097/CCM.0b013e3182a17064. PMID 23989089
- [Background] Balas MC, Vasilevskis EE, Olsen KM, Schmid KK, Shostrom V, Cohen MZ, Peitz G, Gannon DE, Sisson J, Sullivan J, Stothert JC, Lazure J, Nuss SL, Jawa RS, Freihaut F, Ely EW, Burke WJ. Effectiveness and safety of the awakening and breathing coordination, delirium monitoring/management, and early exercise/mobility bundle. Crit Care Med. 2014 May;42(5):1024-36. doi: 10.1097/CCM.0000000000000129. PMID 24394627
- [Background] Skrobik Y, Ahern S, Leblanc M, Marquis F, Awissi DK, Kavanagh BP. Protocolized intensive care unit management of analgesia, sedation, and delirium improves analgesia and subsyndromal delirium rates. Anesth Analg. 2010 Aug;111(2):451-63. doi: 10.1213/ANE.0b013e3181d7e1b8. Epub 2010 Apr 7. PMID 20375300
- [Background] Colombo R, Corona A, Praga F, Minari C, Giannotti C, Castelli A, Raimondi F. A reorientation strategy for reducing delirium in the critically ill. Results of an interventional study. Minerva Anestesiol. 2012 Sep;78(9):1026-33. Epub 2012 Jul 6. PMID 22772860
- [Background] Aghaie B, Rejeh N, Heravi-Karimooi M, Ebadi A, Moradian ST, Vaismoradi M, Jasper M. Effect of nature-based sound therapy on agitation and anxiety in coronary artery bypass graft patients during the weaning of mechanical ventilation: A randomised clinical trial. Int J Nurs Stud. 2014 Apr;51(4):526-38. doi: 10.1016/j.ijnurstu.2013.08.003. Epub 2013 Aug 29. PMID 24035670
- [Background] Hager DN, Dinglas VD, Subhas S, Rowden AM, Neufeld KJ, Bienvenu OJ, Touradji P, Colantuoni E, Reddy DR, Brower RG, Needham DM. Reducing deep sedation and delirium in acute lung injury patients: a quality improvement project. Crit Care Med. 2013 Jun;41(6):1435-42. doi: 10.1097/CCM.0b013e31827ca949. PMID 23507716
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Fan E. Critical illness neuromyopathy and the role of physical therapy and rehabilitation in critically ill patients. Respir Care. 2012 Jun;57(6):933-44; discussion 944-6. doi: 10.4187/respcare.01634. PMID 22663968
- [Background] Collinsworth AW, Priest EL, Campbell CR, Vasilevskis EE, Masica AL. A Review of Multifaceted Care Approaches for the Prevention and Mitigation of Delirium in Intensive Care Units. J Intensive Care Med. 2016 Feb;31(2):127-41. doi: 10.1177/0885066614553925. Epub 2014 Oct 27. PMID 25348864
- [Background] Gerovasili V, Stefanidis K, Vitzilaios K, Karatzanos E, Politis P, Koroneos A, Chatzimichail A, Routsi C, Roussos C, Nanas S. Electrical muscle stimulation preserves the muscle mass of critically ill patients: a randomized study. Crit Care. 2009;13(5):R161. doi: 10.1186/cc8123. Epub 2009 Oct 8. PMID 19814793
- [Background] Gerovasili V, Tripodaki E, Karatzanos E, Pitsolis T, Markaki V, Zervakis D, Routsi C, Roussos C, Nanas S. Short-term systemic effect of electrical muscle stimulation in critically ill patients. Chest. 2009 Nov;136(5):1249-1256. doi: 10.1378/chest.08-2888. Epub 2009 Aug 26. PMID 19710290
- [Background] Morris PE, Griffin L, Berry M, Thompson C, Hite RD, Winkelman C, Hopkins RO, Ross A, Dixon L, Leach S, Haponik E. Receiving early mobility during an intensive care unit admission is a predictor of improved outcomes in acute respiratory failure. Am J Med Sci. 2011 May;341(5):373-7. doi: 10.1097/MAJ.0b013e31820ab4f6. PMID 21358312
- [Background] Cheung AM, Tansey CM, Tomlinson G, Diaz-Granados N, Matte A, Barr A, Mehta S, Mazer CD, Guest CB, Stewart TE, Al-Saidi F, Cooper AB, Cook D, Slutsky AS, Herridge MS. Two-year outcomes, health care use, and costs of survivors of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):538-44. doi: 10.1164/rccm.200505-693OC. Epub 2006 Jun 8. PMID 16763220
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Nordon-Craft A, Schenkman M, Ridgeway K, Benson A, Moss M. Physical therapy management and patient outcomes following ICU-acquired weakness: a case series. J Neurol Phys Ther. 2011 Sep;35(3):133-40. doi: 10.1097/NPT.0b013e3182275905. PMID 21934375
- [Background] Fan E, Cheek F, Chlan L, Gosselink R, Hart N, Herridge MS, Hopkins RO, Hough CL, Kress JP, Latronico N, Moss M, Needham DM, Rich MM, Stevens RD, Wilson KC, Winkelman C, Zochodne DW, Ali NA; ATS Committee on ICU-acquired Weakness in Adults; American Thoracic Society. An official American Thoracic Society Clinical Practice guideline: the diagnosis of intensive care unit-acquired weakness in adults. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1437-46. doi: 10.1164/rccm.201411-2011ST. PMID 25496103
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Adler J, Malone D. Early mobilization in the intensive care unit: a systematic review. Cardiopulm Phys Ther J. 2012 Mar;23(1):5-13. PMID 22807649
- [Background] Elliott D, McKinley S, Alison J, Aitken LM, King M, Leslie GD, Kenny P, Taylor P, Foley R, Burmeister E. Health-related quality of life and physical recovery after a critical illness: a multi-centre randomised controlled trial of a home-based physical rehabilitation program. Crit Care. 2011 Jun 9;15(3):R142. doi: 10.1186/cc10265. PMID 21658221